CLINICAL TRIAL: NCT05014711
Title: Compare the Effects of Remifentanil and Fentanyl on the Duration of Mechanical Ventilation of ICU Patients: a Multi-centre, Randomized, Controlled Trial
Brief Title: Compare the Effects of Remifentanil and Fentanyl on the Duration of Mechanical Ventilation of ICU Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2019-082-02
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Mechanical Ventilation
Keywords: mechanical ventilation; remifentanil; fentanyl; analgesia
MeSH Terms: conditions — Agnosia | interventions — Remifentanil; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remifentanil group (Experimental): After enrollment, remifentanil will be used for analgesia. Duration of mechanical ventilation, incidences of adverse events, interval from SBT to extubation, dosages and costs of analgesics and sedatives drugs will be observed.
  Interventions: Drug: Remifentanil
- fentanil group (Active Comparator): After enrollment, fentanil will be used for analgesia. Duration of mechanical ventilation, incidences of adverse events, interval from SBT to extubation, dosages and costs of analgesics and sedatives drugs will be observed.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Remifentanil — Before infusion, remifentanil is given 0.3 g/kg slowly intravenous injection more than 60 seconds, and the initial dose is 0.025ug/kg/min. The dosage is adjusted to achieve the target depth of analgesia and sedation (CPOT < 3, RASS -2 to 1), with each change 0.025ug/kg/min and the maximum dose 0.15ug/kg/min.
  Other Names: remifentanil hydrochloride
  Arms: remifentanil group
Drug: Fentanyl — Before infusion, fentanyl is given 0.3 g/kg slowly intravenous injection more than 60 seconds, and the initial dose is 0.025ug/kg/min. The dosage is adjusted to achieve the target depth of analgesia and sedation (CPOT < 3, RASS -2 to 1), with each change 0.025ug/kg/min and the maximum dose 0.15ug/kg/min.
  Other Names: Fentanyl citrate
  Arms: fentanil group

SUMMARY:
To verify whether remifentanil is more beneficial to reduce the duration of mechanical ventilation, shorten the interval from SBT to extubation, reduce the incidence of adverse events, reduce the workload of nursing staff, reduce the dosage of sedatives and ICU hospitalization costs, shorten the length of ICU hospitalization, and reduce the short-term mortality.

DETAILED DESCRIPTION:
Opioids are widely used for analgesia in the ICU, of which, fentanyl and remifentanil are the most commonly used. Compared with the two analgesics, fentanyl is relatively cheap, but it is metabolised by liver. Long-term infusion makes its half-life extended, and side effects increase significantly. Respiratory depression is the most serious side effect and may lead to re-intubation and even sudden death.

Remifentanil is a strong selective μ-opioid receptor agonist, rapidly metabolized by non-specific plasma and tissue esterases into inactive metabolites; it has very short context-sensitive half-life even after prolonged infusion or in patients with organ failure. Remifentanil is easy to titrate and provides excellent analgesia: it allows higher doses administration than are normally used with traditional opioids without concerns about accumulation or delayed recovery.

This feature is helpful for patients with mechanical ventilation to weaning and extubate early. Previous studies comparing the two drugs mainly focus on short-term postoperative application, and theoretically long-term use can better reflect the pharmacokinetic advantages of Remifentanil. So we designed this study.

ELIGIBILITY:
Inclusion Criteria:

* (1) Oral endotracheal intubation requiring mechanical ventilation; and (2) 18-85 years old; and (3) expected to require mechanical ventilation for longer than 24 hours.

Exclusion Criteria:

* (1) Deep sedation is required (PaO2/FiO2 ≤100, loss of consciousness during treatment with muscle relaxants, status epilepticus, surgery or surgical conditions require absolute immobilization, severe brain injury with intracranial hypertension, therapeutic hypothermia, etc. And other clinical assessments need to maintain RASS<-2); (2) The time of using sedatives or opioid analgesics is longer than 1 week before enrollment; (3) ICU stay ≥ 1 week before enrollment; (4) Invasive mechanical ventilation time ≥ 48 hours before enrollment; (5) According to the condition of the disease, it is estimated that mechanical ventilation will be needed for too long, such as the accumulation of respiratory muscles in peripheral neuromuscular diseases, brainstem damage and respiratory center involvement; (6) Delirium, alcohol withdrawal symptoms or mental illness or use of antipsychotic drugs; (7) Severe abnormal liver function (Child-Pugh grade C); (8) Renal insufficiency requires renal replacement therapy; (9) Surgical treatment is required during mechanical ventilation (except for minor operations, such as lumbar puncture, ventricular drainage, etc.); (10) Allergy to study drugs or other contraindications; (11) Pregnant or lactating women; (12) Has been selected for other RCT tests; (13) The patient or the legally authorized person is unwilling to participate in the trial; (14) The investigator judged that the patient was not suitable for selection (such as severe hypotension; potential disputes, etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
duration of mechanical ventilation | the end point of time is successfully transferred out of ICU or death or 28 days after enrollment
  from the time of enrollment to successful removal from the ventilator

SECONDARY OUTCOMES:
Incidences of adverse events | 1) Tracheal intubation has been successfully removed; 2) Tracheal intubation has not been removed 15 days after inclusion, and the patient would be followed up for 15 days; 3) Tracheotomy and the ventilator successfully removed,whichever comes first.
  delirium, severe hypotension, severe bradycardia, constipation, chills, nausea and vomiting, muscle rigidity, accidental extubation
the interval from SBT(Spontaneous Breathing Trial) to extubation | the end point of time is successfully transferred out of ICU or death or 28 days after enrollment
  tracheal intubation has been successfully removed after the first SBT
dosages and costs of analgesic and sedative drugs | 1) Tracheal intubation has been successfully removed; 2) Tracheal intubation has not been removed 15 days after inclusion, and the patient would be followed up for 15 days; 3) Tracheotomy and the ventilator successfully removed,whichever comes first.
  The consumption and cost of analgesic and sedative drugs in experimental group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Capital Medical University
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No